CLINICAL TRIAL: NCT02296918
Title: A Phase 1b Study of ACP-196 in Combination With Obinutuzumab for Patients With Relapsed / Refractory or Untreated CLL/SLL/PLL
Brief Title: Acalabrutinib in Combination With Anti-CD20 and Venetoclax in Relapsed/Refractory or Untreated CLL/SLL/PLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-CL-003
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Prolymphocytic Leukemia
Keywords: CLL; SLL; PLL; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Prolymphocytic Leukemia; ACP-196; acalabrutinib; obinutuzumab; rituximab; venetoclax
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — acalabrutinib; obinutuzumab; venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: Acalabrutinib+Obinutuzumab (R/R) (Experimental): Dose-escalation and dose-expansion phases will be conducted for relapsed/refractory (R/R) participants with CLL. In dose-escalation phase, participants will receive oral acalabrutinib Dose 1 once daily (QD), later the dose was switched to Dose 2 twice daily (BID) per Amendment 02. In dose- expansion phase, participants will receive oral acalabrutinib Dose 2 BID in 28-day continuous cycles; and will receive intravenous (IV) infusion of obinutuzumab for total 6 cycles (from Cycles 2 to 7) as on Cycle 2 Day 1 participants will receive Dose 1, on Cycle 2 Day 2 participants will receive Dose 2, on Cycle 2 Days 8 and 15 participants will receive Dose 3, and on Day 1 of Cycles 3 to 7 participants will receive Dose 3. Participants will continue to receive acalabrutinib Dose 2 BID until disease progression, an unacceptable drug-related toxicity, or per the investigator the study treatment is intolerable or no longer in participant's best interest, whichever occurs first.
  Interventions: Drug: acalabrutinib; Drug: Obinutuzumab
- Cohort 2: Acalabrutinib+Obinutuzumab (Treatment-naive) (Experimental): Dose-escalation and dose-expansion phases will be conducted for treatment-naïve participants with CLL/ small lymphocytic lymphoma (SLL). In dose-escalation phase, participants will receive oral acalabrutinib Dose 2 BID in first cycle (28-day cycle). In dose- expansion phase, participants will receive oral acalabrutinib Dose 2 BID in 28-day continuous cycles; and will receive IV infusion of obinutuzumab for total 6 cycles (from Cycles 2 to 7) as on Cycle 2 Day 1 participants will receive Dose 1, on Cycle 2 Day 2 participants will receive Dose 2, on Cycle 2 Days 8 and 15 participants will receive Dose 3, and on Day 1 of Cycles 3 to 7 participants will receive Dose 3. Participants will continue to receive acalabrutinib Dose 2 BID until disease progression, an unacceptable drug-related toxicity, or per the investigator the study treatment is intolerable or no longer in participant's best interest, whichever occurs first.
  Interventions: Drug: acalabrutinib; Drug: Obinutuzumab
- Cohort 3: Acalabrutinib+Rituximab+Venetoclax (R/R) (Experimental): The R/R participants with CLL will receive oral acalabrutinib, IV infusion of rituximab, and oral venetoclax. Participants will receive acalabrutinib Dose 2 BID in 28-day continuous cycles until disease progression, an unacceptable drug-related toxicity, or per the investigator the study treatment is intolerable or no longer in participant's best interest, whichever occurs first. Participants will receive rituximab for total 6 cycles (from Cycles 2 to 7) as Dose 1 on Cycle 2 Day 1, followed by Dose 1 every 3 weeks (Q3W) for 3 doses, then every 4 weeks (Q4W) for 5 doses (total 9 infusions through the end of Cycle 7). Participants will receive venetoclax weekly ramp-up schedule over 5 weeks from Cycles 3 to 15, Dose 1 QD for 1 week on Cycle 3 Day 1, Dose 2 QD for 1 week on Cycle 3 Day 8, Dose 3 QD for 1 week on Cycle 3 Day 15, Dose 4 QD for 1 week on Cycle 3 Day 22, and Dose 5 QD from Cycle 4 Day 1 until completion of Cycle 15.
  Interventions: Drug: acalabrutinib; Drug: Venetoclax; Drug: Rituximab
- Cohort 4: Acalabrutinib+Obinutuzumab+Venetoclax (Treatment-naive) (Experimental): The treatment-naïve participants with CLL will receive oral acalabrutinib, IV infusion of obinutuzumab, and oral venetoclax. Participants will receive acalabrutinib Dose 2 BID in 28-day continuous cycles until disease progression, an unacceptable drug-related toxicity, or per the investigator the study treatment is intolerable or no longer in participant's best interest, whichever occurs first. Participants will receive obinutuzumab for total 6 cycles (from Cycles 2 to 7) as Dose 1 on Cycle 2 Day 1, Dose 2 on Cycle 2 Day 2, Dose 3 on Cycle 2 Days 8 and 15, and Dose 3 on Day 1 of Cycles 3 to 7. Participants will receive venetoclax weekly ramp-up schedule over 5 weeks from Cycles 3 to 15 as Dose 1 QD for 1 week on Cycle 3 Day 1, Dose 2 QD for 1 week on Cycle 3 Day 8, Dose 3 QD for 1 week on Cycle 3 Day 15, Dose 4 QD for 1 week on Cycle 3 Day 22, and from Cycle 4 Day 1 participants will receive Dose 5 QD until completion of Cycle 15.
  Interventions: Drug: acalabrutinib; Drug: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: acalabrutinib — Participants will receive oral acalabrutinib in Cohorts 1, 2, 3, and 4. The details are mentioned in the cohort description.
  Other Names: ACP-196
Drug: Obinutuzumab — Participants will receive intravenous obinutuzumab in Cohorts 1, 2, and 4. The details are mentioned in the cohort description.
  Other Names: Gazyvaro
  Arms: Cohort 1: Acalabrutinib+Obinutuzumab (R/R); Cohort 2: Acalabrutinib+Obinutuzumab (Treatment-naive); Cohort 4: Acalabrutinib+Obinutuzumab+Venetoclax (Treatment-naive)
Drug: Venetoclax — Participants will receive oral venetoclax in Cohorts 3 and 4. The details are mentioned in the cohort description.
  Other Names: ABT-199; Venclexta; GDC-0199
  Arms: Cohort 3: Acalabrutinib+Rituximab+Venetoclax (R/R); Cohort 4: Acalabrutinib+Obinutuzumab+Venetoclax (Treatment-naive)
Drug: Rituximab — Participants will receive intravenous rituximab in Cohort 3. The details are mentioned in the cohort description.
  Other Names: Rituxan
  Arms: Cohort 3: Acalabrutinib+Rituximab+Venetoclax (R/R)

SUMMARY:
To evaluate the safety and preliminary efficacy of acalabrutinib in combination with obinutuzumab in 4 separate cohorts of participants.

DETAILED DESCRIPTION:
A Phase 1b Study of ACP-196 in Combination with Obinutuzumab for Participants with Relapsed/Refractory or Untreated chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL)/ prolymphocytic leukemia (PLL).

Study started with two cohorts, on Acalabrutinib and Obinutuzumab, cohort 1 for relapsed or refractory participants and cohort 2 for treatment naïve participants. Then for longer survival data and combination therapy, two new cohorts added to the study, cohort 3 with relapsed or refractory participants on Acalabrutinib, Rituximab and Venetoclax, and cohort 4 with treatment naïve participants on Acalabrutinib, Obinutuzumab and Venetoclax.

Primary endpoints: For Cohorts 1 and 2, the ORR (PR or better) at the 12-month response assessment will be calculated and 95% exact binomial confidence interval (CIs) will be provided. For Cohorts 1 to 4, toxicities will be tabulated by type and grade using NCI-CTCAE (National Cancer Institute - Common Terminology Criteria for Adverse Events) version 4.03 criteria or higher and displayed in summary form.

Currently, study is in maintenance phase and we don't expect a major change in the near future.

ELIGIBILITY:
Inclusion Criteria

1. Participants with a diagnosis of intermediate or high risk CLL (or variant immunophenotype), SLL, or B-cell prolymphocytic leukemia (B-PLL) by International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria (Hallek et al. 2008) who have:

   * Cohorts 1 and 3: Previously received at least 1 therapy for their disease (Cohort 3 enrollment limited to CLL).
   * Cohort 2: Previously untreated disease and ≥65 years old OR under 65 years old and refuse or are ineligible for chemoimmunotherapy.
   * Cohort 4: Previously untreated disease; Cohort 4 enrollment limited to CLL.
2. Participants in Cohorts 1 and 3 may have received previous ibrutinib (or another Bruton tyrosine kinase (BTK) inhibitor) as long as discontinuation was for a reason other than on-treatment disease progression.
3. All participants must satisfy one of the following criteria for active disease requiring therapy:

   * Evidence of marrow failure as manifested by the development or worsening of anemia or thrombocytopenia (not attributable to autoimmune hemolytic anemia (AIHA) or thrombocytopenia)
   * Massive (≥6 cm below the costal margin), progressive or symptomatic splenomegaly
   * Massive nodes (≥10 cm) or progressive or symptomatic lymphadenopathy
   * Constitutional symptoms, which include any of the following:

   Unintentional weight loss of 10% or more within 6 months Significant fatigue limiting activity Fevers ≥100.5°F for 2 weeks or more without evidence of infection Night sweats >1 month without evidence of infection
4. This criterion was removed with Amendment 5.
5. Participants with a history of Richter's syndrome are eligible if they now have evidence of CLL only, with <10% large cells in the bone marrow.
6. Participants must have adequate organ function, defined as creatinine ≤2.5 times the upper limit of normal range (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x ULN, and bilirubin ≤2.5 x ULN. For Cohorts 3 and 4, participants must have creatinine clearance ≥50 mL/min using modified Cockcroft-Gault equation (using Ideal Body Mass [IBM] instead of mass):
7. IBM (kg) = [(height cm - 154) ● 0.9] + (50 if male, 45.5 if female).
8. Platelets >50 x 10^9/L. In participants with CLL involvement of the marrow, >30 x 10^9/L for Cohorts 1 and 2. For Cohorts 3 and 4, participants must have hemoglobin >9 g/dL.
9. Absolute neutrophil count (ANC) ≥750/mm^3. In participants with CLL involvement of the marrow, ANC ≥500/mm^3. For Cohorts 3 and 4, participants must have ANC ≥1000/mm^3.
10. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
11. Participant must not have secondary cancers that result in a life expectancy of <2 years or that would confound assessment of toxicity in this study.
12. Participants must be ≥18 years of age.
13. Participant must provide written informed consent. A signed copy of the consent form will be retained in the participant's chart.
14. Participant must be able to receive outpatient treatment and follow-up at the treating institution.
15. Participant must have completed all CLL therapies ≥4 weeks prior to first study dose. Palliative steroids are allowed but must be at a dose equivalent of ≤20 mg prednisone daily for at least 1 week prior to treatment initiation.
16. Women who are sexually active and can bear children must agree to use highly effective forms of contraception while on the study and for 2 days after the last dose of acalabrutinib, 30 days after the last dose of venetoclax, 12 months the last dose of rituximab, or 18 months after the last dose of obinutuzumab, whichever is the longest period following the participant's study drug discontinuation. Men who are sexually active and able to have children must agree to use highly effective methods of contraception during the study and use a barrier method (condom; even if the participant had a vasectomy) for 2 days after the last dose of acalabrutinib, 18 months after the last dose of obinutuzumab, or 12 months after the last dose of rituximab, or 30 days after the last dose of venetoclax, whichever is longer. Highly effective forms of contraception are defined in Section 6.4.3. Additionally, men must agree to refrain from sperm donation during the study and for 18 months after the last dose of obinutuzumab, or 12 months after the last dose of rituximab, or 30 days after the last dose of venetoclax, whichever is longer.
17. Participants must be able to swallow whole capsules.
18. Inclusion of women and minorities: Participants of both genders and all racial/ethnic groups are eligible for the study if they meet eligibility criteria outlined. To date, there is no information that suggests that differences in drug metabolism or disease response would be expected in one group compared with another. The small number of participants in a Phase 1b trial precludes any analysis of data to compare participant subgroups based on gender or race/ethnicity.

Exclusion Criteria

1. For Cohorts 2 and 4, received previous therapy for CLL. Treatment of autoimmune complications of CLL with steroids or rituximab is allowed, however, CD20 must have returned on 10% of the CLL cells if rituximab was recently administered. Palliative steroids are acceptable at doses ≤20 mg prednisone equivalent daily.
2. Any life-threatening illness, medical condition, or organ dysfunction, which in the investigator's opinion, could compromise the participants' safety, interfere with the absorption or metabolism of acalabrutinib, or put the study outcomes at undue risk.
3. Female participants who are pregnant or breastfeeding.
4. Participants with active cardiovascular disease not medically controlled or those who have had myocardial infarction in the past 6 months, or corrected QT interval (QTc) ≥480 ms.
5. Malabsorption syndrome, disease significantly affecting gastrointestinal (GI) function, or resection of the stomach or small bowel or gastric bypass, ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
6. Grade >=2 toxicity (other than alopecia) continuing from prior anticancer therapy including radiation.
7. Major surgery within 4 weeks before first dose of study drug.
8. History of a bleeding diathesis (e.g., hemophilia, Von Willebrand disease).
9. Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenia purpura.
10. History of stroke or intracranial hemorrhage within 6 months before the first dose of study drug.
11. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 28 days of first dose of study drug.
12. Requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole).
13. Participants with active infections requiring IV antibiotic/antiviral therapy are not eligible for entry onto the study until resolution of the infection. Participants on prophylactic antibiotics or antivirals are acceptable.
14. Participants with history of or ongoing drug-induced pneumonitis.
15. Participants with human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) or any uncontrolled active systemic infection.
16. Serologic status reflecting active hepatitis B or C infection.

    1. Participants who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative hepatitis B DNA result by polymerase chain reaction (PCR) before randomization. Those who are HBsAg-positive and/or hepatitis B PCR positive will be excluded.
    2. Participants receiving prophylactic intravenous immunoglobulin (IVIG) may have positive hepatitis serologies. Participants who are on IVIG who have positive hepatitis serologies must have a negative hepatitis B DNA to be eligible.
    3. Participants with a history of HBV infection but negative HBV serologies at screening must also have a negative HBV PCR to be eligible.
    4. Participants with a known history of hepatitis C or who are hepatitis C antibody positive should be tested for HCV RNA during screening. Participants who are hepatitis C antibody positive will need to have a negative PCR result before randomization. Those who are hepatitis C PCR positive will be excluded. No further testing beyond screening is necessary if PCR results are negative. However, in the setting of rising transaminase and/or bilirubin levels, HCV PCR testing should be performed when clinically indicated.
17. Participants with substance abuse or other medical or psychiatric conditions that, in the opinion of the investigator, would confound study interpretation or affect the participant's ability to tolerate or complete the study.
18. Participants cannot concurrently participate in another therapeutic clinical trial.
19. Participants who have received a live virus vaccination within 1 month of starting study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Objective Response (OR) at 12 Months as Assessed by the Investigator in Cohorts 1 and 2 | Day 1 through 12 months
  The OR is complete remission (CR), incomplete CR (CRi), nodular partial remission (nPR), or partial remission (PR) for at least 2 months. For CLL, CR:lymphocytes (lympho) <4×10^9/L, normocellular bone marrow (BM) <30% lympho, no B-lymphoid nodules, normal lymph nodes (NLN), liver and spleen (L/S), absolute neutrophils (ANC) >1.5×10^9/L, platelets >100×10^9/L, hemoglobin (Hb) >11g/dL; CRi: lympho <4×10^9/L, hypocellular BM, NLN, L/S, persistent anemia/thrombocytopenia/neutropenia; nPR: CR with present lymphoid nodules (NL); PR: >=50% reduction in lymphadenopathy and/or enlargement of L/S or lympho (<5×10^9/L or >=50% decrease from baseline), criteria of ANC/platelets/Hb per CR or >=50% improvement over baseline. Hematology without exogenous growth factors/transfusion. For SLL, CR: no disease/disease-related symptoms, normal/<=1cm LN, no enlargement of L/S/NL, disease-free BM; PR: >=50% decrease in dominant masses with no size increase/new lesions, and >=50% reduction of nodules in S/L.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Treatment-Emergent Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4 Abnormalities in Laboratory Parameters in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  Participants with treatment-emergent CTCAE Grade 3 or 4 abnormalities in laboratory parameters are reported. Laboratory analysis included hematology, clinical chemistry, and immunology.
Number of Participants With Abnormal Vital Signs Reported as TEAEs in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  Participants with abnormal vital signs (blood pressure, respiratory rate, heart rate, temperature, and body weight) reported as TEAEs are reported.
Number of Participants with Shift From Baseline to Worst (Grade 3 and 4) Post-baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status in all Cohorts | Baseline (Days -28 to -1) through the final data cutoff date (approximately 6 years 8 months)
  The ECOG Performance Status assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=death. Shift from baseline (Days -28 to -1) to worst Grade 3 and/4 in EOCG status are reported.

SECONDARY OUTCOMES:
Percentage of Participants with CR as Assessed by the Investigator in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  For CLL, CR: lymphocytes < 4×10^9/L, normocellular bone marrow < 30% lymphocytes, no B-lymphoid nodules, normal lymph nodes, liver and spleen, absolute neutrophils > 1.5×10^9/L, platelets > 100×10^9/L, hemoglobin > 11g/dL. Hematology without exogenous growth factors/ transfusion. For SLL, CR: no disease/disease-related symptoms, normal/<=1 cm lymph nodes, no enlargement of liver/spleen/lymphoid nodules, disease-free bone marrow.
Percentage of Participants With Minimal Residual Disease (MRD)-negative CR as Assessed by the Investigator in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  For CLL, CR: lymphocytes <4×10^9/L, normocellular bone marrow (BM) <30% lymphocytes, no B-lymphoid nodules, normal lymph nodes, liver, and spleen, absolute neutrophil count >1.5×10^9/L, platelets >100×10^9/L, hemoglobin > 11g/dL; CRi: lymphocytes < 4×10^9/L, hypocellular BM, normal lymph nodes, liver, and spleen, persistent anemia/thrombocytopenia/neutropenia. Hematology without exogenous growth factors/transfusion. For SLL, CR: no disease/disease-related symptoms, normal/<=1 cm lymph nodes, no enlargement of liver/spleen/lymphoid nodules, disease-free BM. MRD negativity was determined in bone marrow by flow cytometry.
Percentage of Participants With OR at Cycle 16 as Assessed by the Investigator in Cohorts 3 and 4 | Day 1 to the end of Cycle 16 (each cycle is 28 days)
  The OR is complete remission (CR), incomplete CR (CRi), nodular partial remission (nPR), or partial remission (PR) for at least 2 months. For CLL, CR: lymphocytes <4×10^9/L, normocellular bone marrow <30% lymphocytes, no B-lymphoid nodules, normal lymph nodes (NLN), liver and spleen (L/S), absolute neutrophils (ANC) >1.5×10^9/L, platelets >100×10^9/L, hemoglobin (Hb) >11g/dL; CRi: lymphocytes <4×10^9/L, hypocellular bone marrow, NLN, L/S, persistent anemia/thrombocytopenia/neutropenia; nPR: CR with present lymphoid nodules; PR: >=50% reduction in lymphadenopathy and/or enlargement of L/S or lymphocytes (<5×10^9/L or >=50% decrease from baseline), criteria of ANC/platelets/Hb per CR or >=50% improvement over baseline. Hematology without exogenous growth factors/transfusion.
Duration of Response (DoR) as Assessed by the Investigator in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  The DoR is defined as the time from the date of achieving the first CR, CRi, nPR, or PR (PR or better) to the date of progressive disease (PD) or death due to any cause, whichever occurred first. The CR, CRi, nPR, and PR are defined in the above outcome measure. For CLL, PD is defined as any one of the criteria: lymphocytes >=50% increase from baseline, appearance of any new lesion or new hepatomegaly or splenomegaly or >= 50% increase in lymphadenopathy/hepatomegaly/splenomegaly, decrease of Hb levels >2 g/dL or to <10 g/dL, or decrease of platelets >50% or to<100,000/μL. For SLL, PD is defined as any one of the criteria: appearance of a new lesion >1.5 cm in any axis; >=50% increase in the products of at least 2 LNs; >=50% increase in the longest diameter of a previously identified node >1 cm in short axis; >=50% increase in the size of the L and/or S or previously determined nodules in the L/S; or new or recurrent BM involvement. The DoR was estimated using Kaplan-Meier method.
Progression Free Survival (PFS) as Assessed by the Investigator in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  The PFS is defined as the time from the date of first dose of study drug to the date of first PD or death due to any cause, whichever occurred first. For CLL, PD is defined as any one of the criteria as: lymphocytes >=50% increase from baseline, appearance of any new lesion or new appearance of hepatomegaly or splenomegaly or >= 50% increase in lymphadenopathy/hepatomegaly/splenomegaly, decrease of Hb levels >2 g/dL or to <10 g/dL, or decrease of platelets >50% or to<100,000/μL. For SLL, PD is defined as any one of the criteria as: appearance of a new lesion >1.5 cm in any axis; >=50% increase in the products of at least 2 LNs; >=50% increase in the longest diameter of a previously identified node >1 cm in short axis; >=50% increase in the size of the L and/or S or previously determined nodules in the L/S; or new or recurrent BM involvement. The PFS was estimated using Kaplan-Meier method.
Time to Next Treatment (TTNT) as Assessed by the Investigator in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  The TTNT is defined as the time from the date of first dose of study drug to the date of institution of subsequent anticancer therapy for CLL or death due to any cause, whichever occurred first. The TTNT was estimated using Kaplan-Meier method.
Overall Survival (OS) as Assessed by the Investigator in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  The OS is defined as the time from the date of first dose of study drug to death due to any cause or last follow-up. The OS was estimated using Kaplan-Meier method.
Time to Initial PR or Better Response as Assessed by the Investigator in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  The time to initial PR or better response is defined as the time from the date of first dose of study drug to the date of first PR or better (ie, CRi or CR). For CLL, CR: lymphocytes (lympho) <4×10^9/L, normocellular bone marrow (BM) <30% lympho, no B-lymphoid nodules, normal lymph nodes (NLN), liver and spleen (L/S), absolute neutrophils (ANC) >1.5×10^9/L, platelets >100×10^9/L, hemoglobin (Hb) >11g/dL; CRi: lympho <4×10^9/L, hypocellular BM, NLN, L/S, persistent anemia/thrombocytopenia/neutropenia; PR: >=50% reduction in lymphadenopathy and/or enlargement of L/S or lympho (<5×10^9/L or >=50% decrease from baseline), criteria of ANC/platelets/Hb per CR or >=50% improvement over baseline. Hematology without exogenous growth factors/transfusion. For SLL, CR: no disease/disease-related symptoms, normal/<=1cm LN, no enlargement of L/S/NL, disease-free BM; PR: >=50% decrease in dominant masses with no size increase/new lesions, and >=50% reduction of nodules in S/L.
Time to Initial CR as Assessed by the Investigator in all Cohorts | Day 1 through the final data cutoff date (approximately 6 years 8 months)
  The time to initial CR is defined as the time from the date of first dose of study drug to the date of first CR. For CLL, CR: lymphocytes < 4×10^9/L, normocellular bone marrow < 30% lymphocytes, no B-lymphoid nodules, normal lymph nodes, liver and spleen, absolute neutrophils > 1.5×10^9/L, platelets > 100×10^9/L, hemoglobin > 11g/dL. Hematology without exogenous growth factors/ transfusion. For SLL, CR: no disease/disease-related symptoms, normal/<=1 cm lymph nodes, no enlargement of liver/spleen/lymphoid nodules, disease-free bone marrow.
Time of Maximum Plasma Concentration (Tmax) of Acalabrutinib and its Metabolite ACP-5862 in Cohorts 1, 3, and 4 | During Cohort 1: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycle 1. Cohorts 3 and 4: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycles 1, 3, and 5. (each cycle is 28 days)
  The Tmax of acalabrutinib and its metabolite ACP-5862 are reported.
Time of Maximum Plasma Concentration (Tmax) of Venetoclax in Cohorts 3 and 4 | Predose and at 0.5, 1, 2, 3, 4, 6, and 24 hours post dose on Cycle 3 Day 1 and Cycle 5 Day 1. (each cycle is 28 days).
  The Tmax of venetoclax is reported.
Maximum Observed Plasma Concentration (Cmax) of Acalabrutinib and its Metabolite ACP-5862 in Cohorts 1, 3, and 4 | Cohort 1: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycle 1. Cohorts 3 and 4: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycles 1, 3, and 5. (each cycle is 28 days)
  The Cmax of acalabrutinib and ACP-5862 are reported.
Maximum Observed Plasma Concentration (Cmax) of Venetoclax in Cohorts 3 and 4 | Predose and at 0.5, 1, 2, 3, 4, 6, and 24 hours post dose on Cycle 3 Day 1 and Cycle 5 Day 1. (each cycle is 28 days)
  The Cmax of venetoclax is reported.
Area Under the Plasma Concentration-time Curve From Time 0 to 6 Hours (AUC0-6) of Acalabrutinib in Cohort 1 | Pre-dose; 0.5, 1, 2, 3, 4, and 6 hours post-dose for Cycle 1. (each cycle is 28 days)
  The AUC0-6 of acalabrutinib is reported.
Area Under the Plasma Concentration-time Curve From Time 0 to 6 Hours (AUC0-6) of Venetoclax in Cohorts 3 and 4 | Predose and at 0.5, 1, 2, 3, 4, 6, and 24 hours post dose on Cycle 3 Day 1 and Cycle 5 Day 1. (each cycle is 28 days)
  The AUC0-6 of venetoclax is reported.
Area Under the Plasma Concentration-time Curve From Time 0 to Last Measurable Concentration (AUC0-last) of Acalabrutinib and its Metabolite ACP-5862 in Cohorts 1, 3, and 4 | Cohort 1: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycle 1. Cohorts 3 and 4: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycles 1, 3, and 5.(each cycle is 28 days)
  The AUC0-last of acalabrutinib and ACE-5862 are reported.
Area Under the Plasma Concentration-time Curve From Time 0 to Last Measurable Concentration (AUC0-last) of Venetoclax in Cohorts 3 and 4 | Predose and at 0.5, 1, 2, 3, 4, 6, and 24 hours post dose on Cycle 3 Day 1 and Cycle 5 Day 1. (each cycle is 28 days)
  The AUC0-last of venetoclax is reported.
Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to infinity (AUC0-inf) of Acalabrutinib and its Metabolite ACP-5862 in Cohorts 1, 3, and 4 | Cohort 1: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycle 1. Cohorts 3 and 4: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycles 1, 3, and 5. (each cycle is 28 days)
  The AUC0-inf of acalabrutinib and ACE-5862 are reported.
Terminal Elimination Rate Constant (λz) of Acalabrutinib and its Metabolite ACP-5862 in Cohorts 1, 3, and 4 | Cohort 1: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycle 1. Cohorts 3 and 4: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycles 1, 3, and 5. (each cycle is 28 days)
  The λz of acalabrutinib and ACP-5862 are reported.
Apparent oral clearance (CL/F) of Administration of Acalabrutinib in Cohorts 1, 3, and 4 | Cohort 1: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycle 1. Cohorts 3 and 4: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycles 1, 3, and 5. (each cycle is 28 days)
  The CL/F of acalabrutinib is reported.
Apparent Volume of Distribution (Vz/F) of Acalabrutinib in Cohorts 1, 3, and 4 | Cohort 1: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycle 1. Cohorts 3 and 4: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycles 1, 3, and 5. (each cycle is 28 days)
  The Vz/F of acalabrutinib is reported.
Terminal Elimination Half-life (t1/2) of Acalabrutinib and its Metabolite ACP-5862 in Cohorts 1, 3, and 4 | Cohort 1: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycle 1. Cohorts 3 and 4: pre-dose; 0.5, 1, 2, 3, 4, 6, and 24 hours post-dose for Cycles 1, 3, and 5. (each cycle is 28 days)
  The t1/2 of acalabrutinib and ACP-5862 are reported.
The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) Scores in Cohorts 3 and 4 | At the end of Cycle 2 and Cycle 42 (each cycle is 28 days).
  The EORTC QLQ-C30 is a 30-item questionnaire designed to assess health related quality of life in cancer participants. It includes a 30-item questionnaire designed to assess health related quality of life in cancer patients. There are 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 3 symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. Several single-item symptom measures are also included (dyspnea, insomnia, appetite, constipation, diarrhea, and financial impact). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100. A high score for a functional scale represents a high (healthy/better) level of functioning, a high score for the global health status represents a high (better) quality of life, but a high score for a symptom scale represents a high (worse) level of symptoms/problems.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Study Information Center, Study Director — 1-877-240-9479; information.center@astrazeneca.com
Locations (1):
- Research Site, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Result] Woyach JA, Blachly JS, Rogers KA, Bhat SA, Jianfar M, Lozanski G, Weiss DM, Andersen BL, Gulrajani M, Frigault MM, Hamdy A, Izumi R, Munugalavadla V, Quah C, Wang MH, Byrd JC. Acalabrutinib plus Obinutuzumab in Treatment-Naive and Relapsed/Refractory Chronic Lymphocytic Leukemia. Cancer Discov. 2020 Mar;10(3):394-405. doi: 10.1158/2159-8290.CD-19-1130. Epub 2020 Jan 8. PMID 31915195
- [Derived] Arrato NA, Valentine TR, Byrd JC, Jones JA, Maddocks KJ, Woyach JA, Andersen BL. Illness representations and psychological outcomes in chronic lymphocytic leukaemia. Br J Health Psychol. 2022 May;27(2):553-570. doi: 10.1111/bjhp.12562. Epub 2021 Oct 4. PMID 34608724
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-003&attachmentIdentifier=de273ce6-7af3-4729-9533-778cf63bb3af&fileName=ACE-CL-003_CSR_BODY_ace-cl-003_final_CSR_combined-redact.pdf&versionIdentifier=

DOCUMENTS (2):
  • Study Protocol (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT02296918/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT02296918/SAP_001.pdf